CLINICAL TRIAL: NCT01497587
Title: A Single Centre, Open-labelled Trial to Investigate the Pharmacokinetics of Insulin Detemir in Healthy Taiwanese Subjects
Brief Title: Pharmacokinetics of Insulin Detemir in Healthy Volunteers From Taiwan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3023
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin detemir (Experimental)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Single dose, 0.5 U/kg, administered s.c. (under the skin)

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate pharmacokinetics of insulin detemir in healthy Taiwanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination as judged by the investigator
* Body mass index (BMI) between 18 and 27 kg/m^2, inclusive
* Fasting plasma glucose maximum 6.1 mmol/l
* Non-smoker or smoking maximum 5 cigarettes per day or the equivalent

Exclusion Criteria:

* Participation in any other clinical trial involving other investigational products within the last 3 months
* Subject with a history of alcohol or drug dependence
* Subject with a first-degree relative with diabetes mellitus

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Area under the insulin detemir concentration curve

SECONDARY OUTCOMES:
Maximum insulin detemir concentration
Time to maximum insulin detemir concentration
The mean residence time of insulin detemir
Insulin detemir half-life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Taipei, Taiwan

REFERENCES:
- [Result] Kwok C-F, Tsai T-H, Lim S-H, Vaz J, Ho L-T. The Pharmacokinetic Profile of Insulin Detemir in Healthy Male Taiwanese and Caucasian Subjects. ASEAN Federation of Endocrine Societies (AFES); Country: Malaysia City: Kuala Lumpur
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com